CLINICAL TRIAL: NCT05425173
Title: Effect of Limbs Range of Motion Exercises Along With Chest Physical Therapy on Cardiopulmonary Parameters After Correction of Congenital Heart Diseases in ICU
Brief Title: Limbs Range of Motion Exercises Along With Chest Physical Therapy After Correction of Congenital Heart Diseases in ICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Muneeba Gul
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional treatment (Active Comparator): Chest Physical Therapy
  Interventions: Other: Conventional treatment
- Limb Range of Motion Exercises + Chest Physical Therapy (Experimental): Limb Range of Motion Exercises + Chest Physical Therapy
  Interventions: Other: Limb Range of Motion Exercises + Chest Physical Therapy

INTERVENTIONS:
Other: Conventional treatment — Chest Physical Therapy as required
  Arms: Conventional treatment
Other: Limb Range of Motion Exercises + Chest Physical Therapy — Limb Range of Motion Exercises + Chest Physical Therapy
  Frequency: 4 sessions Time: 5 to 10 minutes
  Arms: Limb Range of Motion Exercises + Chest Physical Therapy

SUMMARY:
1. To determine the effect of limb ROMs along with chest Physical therapy on cardiopulmonary parameters after correction of congenital heart diseases in ICU
2. To determine the response of Inotropic drug in relation to Limb ROMs after Correction of Congenital heart diseases in ICU

ELIGIBILITY:
Inclusion Criteria:

* Patients below the age 5 years old that underwent congenital heart surgery.

Exclusion Criteria:

* Contraindications for exercise, mental retardation, unstable hemodynamics

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Heart Rate | Upto 10 days
  Changes from baseline, Heart rate was measured per minute through cardiac monitor
Respiration Rate | Upto 10 days
  Changes from baseline,respiratory rate was measured per minute through cardiac monitor
Systolic Blood Pressure | Upto 10 days
  Changes from the Baseline, Blood pressure is measured through sphygmomanometer
Diastolic Blood Pressure | Upto 10 days
  Changes from the Baseline, Blood pressure is measured through sphygmomanometer
Partial pressure of oxygen | Upto 10 days
  Changes from the Baseline, Blood pressure is measured through sphygmomanometer
Partial Pressure of carbon dioxide | Upto 10 days
  Changes from the Baseline, Blood pressure is measured through sphygmomanometer
Arterial blood gas (ABG) parameter like potential of hydrogen (PH) | Upto 10 days
  Above parameter was measured by serial ABG analysis. Its normal reference range is 7.35-7.45. baseline reading will be taken at 10 minutes before starting Non invasive ventilation training. Changes from the Baseline
Arterial blood gas parameter like bicarbonate(HCO3). | Upto 10 days
  Above parameter was measured by serial ABG analysis. Its normal reference range is 22-28 nmol/L. Baseline reading will be taken at 10 minutes before starting Non invasive ventilation training. Changes from the Baseline
Oxygen saturation | Upto 10 days
  Changes from baseline SPO2 was measured in percentage. Oxygen immersion is the division of oxygen-soaked hemoglobin with respect to add up to hemoglobin in the blood. Pulse oximeter measure it.
Ejection fraction | Upto 10 days
  Change from baseline Ejection fraction through Echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Iqbal Tariq, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Rehman Medical Institute, Peshawar, Khyber PkahtoonKhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No